CLINICAL TRIAL: NCT00510276
Title: A Double-Blind Study of Atomoxetine Hydrochloride Versus Placebo for the Treatment of ADHD in Young Adults With an Assessment of Associated Functional Outcomes
Brief Title: Treatment of Attention-Deficit/Hyperactivity Disorder (ADHD) With Atomoxetine in Young Adults and Its Effects on Functional Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10803; B4Z-US-LYDZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Results first posted 2010-03-03 (Estimated); Last update posted 2010-04-14 (Estimated); Status verified 2010-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental)
  Interventions: Drug: Atomoxetine hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine hydrochloride — 20-50 mg, twice a day per by mouth for 12 weeks, followed by up to an additional 12 weeks
  Other Names: LY139603; Strattera
  Arms: Atomoxetine
Drug: Placebo — twice a day, by mouth for 12 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate atomoxetine's efficacy in treating attention-deficit/hyperactivity disorder (ADHD) symptoms and atomoxetine's effect on functional outcomes in young adults.

A gatekeeper strategy will be employed for sequentially testing the secondary objectives.

This study also has an observational community sample arm in which patients will complete all the efficacy measurements via web-based self reporting.

ELIGIBILITY:
Inclusion Criteria:

* positive attention-deficit/hyperactivity disorder (ADHD) diagnosis with at least moderate severity
* male or female 18 to 30 years of age
* must be able to swallow capsules
* must be able to communicate effectively in English
* must not have cognitive impairment
* be reliable to keep appointments for clinic visits and all related tests

Exclusion Criteria:

* patients diagnosed with obsessive-compulsive disorder, bipolar affective disorder, or psychosis
* females who are pregnant or breastfeeding
* patients with dementia or traumatic brain injury
* patients with a history of severe allergy to atomoxetine
* have untreated hypertension or thyroid problem
* have serious medical illness including any heart, liver, kidney, respiratory, blood, endocrine, or neuromuscular diseases

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 445 (Actual)
Dates: Start 2007-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- United States (27):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rolling Hills Est., California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spring Valley, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wildomar, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagle, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Belmont, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington Hills, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piscataway, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beachwood, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woodstock, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Midlothian, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hato Rey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan

REFERENCES:
- [Derived] Adler LA, Clemow DB, Williams DW, Durell TM. Atomoxetine effects on executive function as measured by the BRIEF--a in young adults with ADHD: a randomized, double-blind, placebo-controlled study. PLoS One. 2014 Aug 22;9(8):e104175. doi: 10.1371/journal.pone.0104175. eCollection 2014. PMID 25148243
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] Durell TM, Adler LA, Williams DW, Deldar A, McGough JJ, Glaser PE, Rubin RL, Pigott TA, Sarkis EH, Fox BK. Atomoxetine treatment of attention-deficit/hyperactivity disorder in young adults with assessment of functional outcomes: a randomized, double-blind, placebo-controlled clinical trial. J Clin Psychopharmacol. 2013 Feb;33(1):45-54. doi: 10.1097/JCP.0b013e31827d8a23. PMID 23277268
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from 16 August 2007 until 19 August 2008 in medical clinics.
Pre-assignment Details: Study Period 1 was a screening/washout period. Subjects who did not meet enrollment criteria were excluded from the trial before randomization. 584 participants entered the screening phase, 139 were screen failures. There was an optional 12-week open-label atomoxetine extension phase after the 12-week acute double-blind phase.
Groups:
- Atomoxetine: 20-50 mg twice a day for 12 weeks, then up to an additional 12 weeks
- Placebo: twice a day for 12 weeks
Period: Acute Double-Blind Phase
Arm/Group | Atomoxetine | Placebo
Started | 220 | 225
Completed | 115 | 130
Not Completed | 105 | 95
Not completed — Adverse Event | 21 | 6
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Lack of Efficacy | 3 | 4
Not completed — Lost to Follow-up | 48 | 49
Not completed — Physician Decision | 0 | 3
Not completed — Protocol Violation | 4 | 3
Not completed — Sponsor Decision | 2 | 1
Not completed — Subject Decision | 26 | 28
Period: Extension Open-Label Phase
Arm/Group | Atomoxetine | Placebo
Started | 111 (4 patients who completed acute phase did not participate in the optional atomoxetine extension phase) | 129 (1 patient who completed acute phase did not participate in the optional atometine extension phase)
Completed | 78 | 81
Not Completed | 33 | 48
Not completed — Adverse Event | 9 | 18
Not completed — Lack of Efficacy | 2 | 7
Not completed — Lost to Follow-up | 12 | 10
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Sponsor Decision | 1 | 0
Not completed — Subject Decision | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atomoxetine | Placebo | Total
Number analyzed (Participants) | 220 | 225 | 445
Age Continuous [Mean (Standard Deviation); unit: years] | 24.71 (3.35) | 24.68 (3.48) | 24.69 (3.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 98 | 190
  Male | 128 | 127 | 255
Region of Enrollment [Number; unit: participants]
  United States | 210 | 220 | 430
  Puerto Rico | 10 | 5 | 15
Adult Attention-Deficit/Hyperactivity Disorder Quality of Life 29 - Life Outlook Subscale [Mean (Standard Deviation); unit: units on a scale] — Patient-reported outcome measure used to examine the disease specific functional impairments and quality of life for adults with ADHD. This subscale assesses life outlook. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
  units on a scale | 54.40 (15.42) | 52.49 (15.41) | 53.44 (15.43)
Adult Attention-Deficit/Hyperactivity Disorder Quality of Life 29 - Psychological Health Subscale [Mean (Standard Deviation); unit: units on a scale] — Patient-reported outcome measure used to examine the disease specific functional impairments and quality of life for adults with ADHD. This subscale assesses the psychological health. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
  units on a scale | 49.89 (18.95) | 50.98 (18.20) | 50.44 (18.56)
Adult Attention-Deficit/Hyperactivity Disorder Quality of Life 29 - Total Score [Mean (Standard Deviation); unit: units on a scale] — Patient-reported outcome measure used to examine the disease-specific functional impariments and quality of life for adults with ADHD. The domains included in the AAQOL are life productivity, psychological health, quality of relationships, and life outlook. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
  units on a scale | 45.95 (13.74) | 45.30 (13.53) | 45.62 (13.62)
Adult Attention-Deficit/Hyperactivity Disorder Quality of Life 29 - relationship subscale [Mean (Standard Deviation); unit: units on a scale] — Patient-reported outcome measure used to examine the disease-specific functional impariments and quality of life for adults with ADHD. This subscale assesses quality of relationships. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
  units on a scale | 52.76 (19.35) | 52.47 (19.67) | 52.61 (19.49)
Beck Anxiety Inventory (BAI) [Mean (Standard Deviation); unit: units on a scale] — 21-item self-reported screening tool for measuring anxiety severity. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely; I could barely stand it). Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety. Patients record how much they have been bothered by each symptom during the past week, including the day the questionnaire is administered. The total score ranges from 0 to 63.
  units on a scale | 10.98 (9.69) | 9.18 (8.47) | 10.07 (9.13)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Behavioral Regulation [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A behavioral regulation subscale measures an individuals control over behavior in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 30 to 90.
  units on a scale | 62.40 (11.91) | 60.94 (10.77) | 61.66 (11.36)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Emotional Control [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A emotional control subscale assesses an individuals emotional control in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 10 to 30.
  units on a scale | 18.76 (5.73) | 18.22 (5.33) | 18.49 (5.53)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - GEC [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Global Executive Composite (GEC) rates the global executive composite of the patient in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 75 to 225.
  units on a scale | 157.11 (22.80) | 156.12 (21.00) | 156.61 (21.89)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Inconsistency [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Inconsistency rates the behavioral inconsistency displayed by the patient in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score is calculated based on a weighted secondary scoring system and ranges from 0 to 20.
  units on a scale | 3.22 (1.86) | 3.50 (1.97) | 3.36 (1.92)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Infrequency [Mean (Standard Deviation); unit: units on a scale] — BRIEF-A Infrequency is a standardized measure assessing adult executive functioning/self-regulation in his/her everyday environment. Extent to which the respondent answers additional items in an unusual and infrequent direction. Self-report form is designed to be completed by adults 18-90 years of age. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. Total score is calculated based on weighted secondary scoring system and ranges from 0 to 5.
  units on a scale | 0.13 (0.40) | 0.15 (0.38) | 0.14 (0.39)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Inhibit [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Inhibit rates an individual's inhibition in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
  units on a scale | 18.28 (2.77) | 18.11 (2.72) | 18.19 (2.74)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Initiate [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Initiate rates an individual's initiative behaviors in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
  units on a scale | 18.33 (3.11) | 18.32 (3.00) | 18.33 (3.05)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Metacognition Index [Mean (Standard Deviation); unit: units on a scale] — BRIEF-A Metacognition subscale is a standardized measure assessing individual's ability to systematically solve problems via planning and organization while sustaining these task-completion efforts in active working memory. Form is designed to be completed by adults, including adults with wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior never observed, 2=behavior sometimes observed, and 3=behavior often observed - higher ratings indicate greater perceived impairment. Total score ranges from 40 to 120.
  units on a scale | 94.71 (13.69) | 95.18 (12.77) | 94.95 (13.22)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Negativity [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Negativity asseses an indivduals' perceived negativity in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score is calculated based on a weighted secondary scoring system and ranges from 0 to 10.
  units on a scale | 2.22 (2.16) | 2.06 (2.03) | 2.14 (2.10)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Plan/Organize [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Plan/Organize asseses an individuals' capabilities to plan and organize in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 10 to 30.
  units on a scale | 23.25 (4.02) | 23.31 (3.91) | 23.28 (3.96)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - SHIFT [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Shift assess an individuals' shifting between different behaviors in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
  units on a scale | 12.56 (2.82) | 12.36 (2.64) | 12.46 (2.73)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Self Monitor [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Self Monitor assesses an individuals' capacity to self monitor in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
  units on a scale | 12.80 (3.01) | 12.25 (2.89) | 12.52 (2.96)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Task Monitor [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Task Monitor assesses an individuals's ability to monitor a task in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
  units on a scale | 14.44 (2.36) | 14.68 (2.31) | 14.56 (2.33)
Behavior Rating Inventory of Executive Function-Adult Version Self Report - Working Memory [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Working Memory assesses an individuals' memory function in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
  units on a scale | 19.87 (2.73) | 19.87 (2.69) | 19.87 (2.71)
Behavior Rating Inventory of Executive Function-Adult Version Self Report- Organization of Materials [Mean (Standard Deviation); unit: units on a scale] — The BRIEF-A Organization of Materials assesses an individuals' organizing skills in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
  units on a scale | 18.82 (4.07) | 19.00 (3.87) | 18.91 (3.97)
Clinical Global Impression-ADHD- Severity (CGI-ADHD-S) [Mean (Standard Deviation); unit: units on a scale] — Single-item clinician rating of the clinician's assessment of the patient's severity of the ADHD symptoms in relation to the clinician's total experience with ADHD patients. Severity is rated on a 7-point scale (1 = normal, not at all ill; 7 = among the most extremely ill patients). The total score ranges from 1 to 7.
  units on a scale | 4.79 (0.66) | 4.68 (0.64) | 4.74 (0.65)
Conners' ADHD Rating Scale Self Report (CAARS-S:SV) Total Score [Mean (Standard Deviation); unit: units on a scale] — The CAARS-S:SV is a 30-item patient-reported scale with 3 subscales: Inattention subscale, Hyperactivity-Impulsivity subscale, and ADHD Index. 18-item total ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each individual item is scored on a 0 to 3 scale (0 = not at all, never; 1 = just a little, once in a while; 2 = Pretty much, often; 3 = very much, very frequently). The rating scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
  units on a scale | 35.01 (8.97) | 35.69 (8.60) | 35.36 (8.78)
Conners' Adult ADHD Rating Scale - Investigator Rated:Screening Version Total Score [Mean (Standard Deviation); unit: units on a scale] — CAARS-Inv:SV is a 30-item scale containing 3 subscales: the Inattention subscale, the Hyperactivity-Impulsivity subscale, and the ADHD Index. The 18-item total ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each item is scored on a 0 to 3 scale (0=not at all, never; 1=just a little, once in a while; 2=pretty much, often; 3=very much, very frequently). The scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
  units on a scale | 39.15 (7.48) | 38.95 (7.72) | 39.05 (7.59)
Driving Behavior Survey Self-Report [Mean (Standard Deviation); unit: units on a scale] — 26 item self-rated driving survey with examples of driving behaviors, e.g.: putting on seat belt, driving within speed limits, yielding the right of way to other drivers. Items are rated on a 4-point scale (1 = not at all or rarely, 2 = sometimes, 3 = often, 4 = very often). The total score is the sum of the 26 items. A driving history is completed by self-report the first time a rater completes the Driving Behavior Survey (Self-Report). The total score ranges from 26 to 104.
  units on a scale | 79.86 (12.89) | 78.95 (12.46) | 79.41 (12.67)
Driving Behavior Survey-Other Report [Mean (Standard Deviation); unit: units on a scale] — 26-item driving survey completed by someone other than the patient/driver. Examples of driving behaviors included in the survey match those listed in the Self-Report version of the scale. Items are rated on a 4-point scale (1 = not at all or rarely, 2 = sometimes, 3 = often, 4 = very often). The total score is the sum of the 26 items and ranges from 26 to 104.
  units on a scale | 70.90 (10.13) | 78.00 (11.24) | 74.77 (11.21)
Epworth Sleepiness Scale (ESS) [Mean (Standard Deviation); unit: units on a scale] — Used to determine the level of daytime sleepiness. The ESS is a self-rated questionnaire with 8 items that describe normative daily situations known to vary in their soporific qualities. Subjects rate the likelihood of dozing off or falling asleep in each of these situations. Each item is rated on a 4-point scale from 0 (would never doze) to 3 (high chance of dozing). The item scores are summed to produce a total score (range of 0-24). Score >10 (95th percentile) are considered to be suggestive of significant daytime sleepiness.
  units on a scale | 9.82 (4.71) | 9.60 (4.74) | 9.71 (4.72)
Fagerstrom Test for Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: units on a scale] — The FTND was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. The FTND contains 4 yes-no and 2 multiple choice questions and can be used in a self-report format. The items on FTND are scored 0 to 3 for multiple choice items, the items are summed to yield a total score of 0-10 (0=minimum nicotine dependence; 10=maximum nicotine dependence).
  units on a scale | 2.08 (2.10) | 2.33 (2.22) | 2.20 (2.16)
Habits Timeline Followback (TLFB) Incidence for Use of Alcohol [Mean (Standard Deviation); unit: number of alcoholic drinks per day] — Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed.
  number of alcoholic drinks per day | 0.98 (1.33) | 1.08 (1.44) | 1.03 (1.38)
Habits Timeline Followback (TLFB) Incidence for Use of Caffeine [Mean (Standard Deviation); unit: number of caffeinated drinks per day] — Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of caffeine consumed by an individual. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome.
  number of caffeinated drinks per day | 1.78 (1.72) | 1.87 (3.19) | 1.82 (2.55)
Habits Timeline Followback (TLFB) Incidence for Use of Drugs [Mean (Standard Deviation); unit: ratio] — Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of recreational drugs other than marijuana an individual consumed and is expressed as the ratio of number of days on which drugs were used over the total number of days, resulting in a total score ranging from 0 to 1. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year.
  ratio | 0.13 (0.15) | 0.27 (0.37) | 0.18 (0.24)
Habits Timeline Followback (TLFB) Incidence for Use of Marijuana [Mean (Standard Deviation); unit: number of joints smoked per day] — Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of marjuana consumed by an individual. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of joints that have been consumed.
  number of joints smoked per day | 0.39 (0.59) | 0.28 (0.38) | 0.34 (0.50)
Habits Timeline Followback (TLFB) Incidence for Use of Nicotine [Mean (Standard Deviation); unit: number of nicotine-products used per day] — Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of nicotine consumed by an individual. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome.
  number of nicotine-products used per day | 6.91 (7.73) | 6.41 (7.44) | 6.65 (7.57)
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] — Rating scale for severity of depressive mood symptoms, administered by the investigator. The scale consists of 10 items, each rated on a scale from 0 to 6. The MADRS total score is the sum of the 10 items and the score ranges from 0 to 60. Higher scores denote more severe depressive symptoms.
  units on a scale | 6.68 (4.28) | 6.29 (4.01) | 6.48 (4.14)
Social Adaptation Self-Evaluation Scale (SASS) [Mean (Standard Deviation); unit: units on a scale] — The SASS is a patient completed scale that consists of 21 items that examine behavior and subjective perception, including satisfaction, self-perception and motivation in participating in and maintaining relationships with family and friends, satisfaction in work, home and leisure activities, and intellectual interests. Each item is scored from 0 to 3, corresponding to minimal and maximal social adjustment, with a total score range from 0 to 60.
  units on a scale | 36.99 (6.17) | 37.28 (5.93) | 37.14 (6.04)

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life-29 (AAQOL-29) Total Score
Description: Patient-reported outcome measure used to examine the disease-specific functional impariments and quality of life for adults with ADHD. The domains included in the AAQOL are life productivity, psychological health, quality of relationships, and life outlook. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
Time Frame: Baseline, 12 weeks
Population: Analyzed was an intent-to-treat population. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 117 | 131
units on a scale | 15.76 (1.28) | 10.95 (1.23)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in AAQOL-29 score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — A gate-keeper strategy was applied to adjust for multiple tests; Mean Difference (Final Values) = 4.82, 95% CI 2-sided [1.44 to 8.20]

2. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life-29 (AAQOL-29) Relationship Subscale
Description: Patient-reported outcome measure used to examine the disease-specific functional impariments and quality of life for adults with ADHD. This subscale asseses quality of relationships. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
Time Frame: Baseline, 12 weeks
Population: Intent-to-treat population was used for analysis. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 117 | 131
units on a scale | 15.51 (1.60) | 9.61 (1.54)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in AAQOL-29 relationship subscale score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis — A gate-keeper strategy was applied to adjust for multiple tests; Mean Difference (Final Values) = 5.90, 95% CI 2-sided [1.68 to 10.12]

3. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life-29 (AAQOL-29) Life Productivity Subscale
Description: Patient-reported outcome measure used to examine the disease specific functional impairments and quality of life for adults with ADHD. This subscale assesses life productivity. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
Time Frame: Baseline, 12 weeks
Population: An intent-to-treat population was analyzed. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 117 | 131
units on a scale | 20.92 (1.79) | 15.18 (1.72)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis — A gate-keeper strategy was applied to adjust for multiple tests; Mean Difference (Final Values) = 5.73, 95% CI 2-sided [1.00 to 10.46]

4. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life-29 (AAQOL-29) Psychological Health Subscale
Description: Patient-reported outcome measure used to examine the disease specific functional impairments and quality of life for adults with ADHD. This subscale asseses the psychological health. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
Time Frame: Baseline, 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 117 | 131
units on a scale | 14.57 (1.53) | 10.21 (1.47)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in AAQOL-29 psychological health subscale score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis — A gate-keeper strategy was applied to adjust for multiple tests; Mean Difference (Final Values) = 4.36, 95% CI 2-sided [0.33 to 8.39]

5. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Quality of Life-29 (AAQOL-29) Life Outlook Subscale
Description: Patient-reported outcome measure used to examine the disease specific functional impairments and quality of life for adults with ADHD. This subscale asseses life outlook. Individual items are scored on a five-point Likert-like scale from "not at all/never=1" to "extremely/very often=5". The range of scores for this subscale is 0 to 100. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
Time Frame: Baseline, 12 weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 117 | 131
units on a scale | 9.27 (1.40) | 5.87 (1.33)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in AAQOL-29 life outlook subscale score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.074, ANCOVA — A gate-keeper strategy was applied to adjust for multiple tests; Mean Difference (Final Values) = 3.40, 95% CI 2-sided [-0.33 to 7.12]

6. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint in Clinical Global Impression-ADHD- Severity (CGI-ADHD-S)
Description: Single-item clinician rating of the clinician's assessment of the patient's severity of the ADHD symptoms in relation to the clinician's total experience with ADHD patients. Severity is rated on a 7-point scale (1 = normal, not at all ill; 7 = among the most extremely ill patients). The total score ranges from 1 to 7.
Time Frame: Baseline, 12 weeks
Population: Analyzed was an intent-to-treat population using last observation carried forward imputation technique. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 192 | 200
units on a scale | -1.10 (0.08) | -0.67 (0.08)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in CGI-ADHD-S score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.63 to -0.24]

7. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint in CAARS Self Report (CAARS-S:SV) Total Score
Description: 30-item patient-reported scale with 3 subscales: Inattention subscale, Hyperactivity-Impulsivity subscale, and ADHD Index. 18-item total ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each individual item is scored on a 0 to 3 scale (0 = not at all, never; 1 = just a little, once in a while; 2 = Pretty much, often; 3 = very much, very frequently). The rating scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
Time Frame: Baseline, 12 weeks
Population: An intent-to-treat population was analyzed using last observation carried forward imputation technique. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 189 | 197
units on a scale | -11.88 (0.75) | -7.84 (0.73)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in CAARS-S:SV score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.04, 95% CI 2-sided [-5.94 to -2.15]

8. Secondary Outcome: Endpoint Scores in Patient Global Impression - Improvement (PGI-I)
Description: 7-point scale modeled after the CGI on which patients rate any change in their overall status that they had experienced since beginning the study drug. The score on this scale ranges from 1 (very much improved) to 7 (very much worse).
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 189 | 197
units on a scale | 3.17 (0.08) | 3.42 (0.08)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in PGI-I scores at 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.020, ANCOVA; ANCOVA with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.45 to -0.04]

9. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Montgomery Asberg Depression Rating Scale (MADRS)
Description: Rating scale for severity of depressive mood symptoms, administered by the investigator. The scale consists of 10 items, each rated on a scale from 0 to 6. The MADRS total score is the sum of the 10 items and the score ranges from 0 to 60. Higher scores denote more severe depressive symptoms.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 173 | 177
units on a scale | -0.72 (0.30) | -0.30 (0.30)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in MADRS score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.282, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-1.19 to 0.35]

10. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Beck Anxiety Inventory (BAI)
Description: 21-item self-reported screening tool for measuring anxiety severity. Each item is rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (severely; I could barely stand it). Each item is descriptive of subjective, somatic, or panic-related symptoms of anxiety. Patients record how much they have been bothered by each symptom during the past week, including the day the questionnaire is administered. The total score ranges from 0 to 63.
Time Frame: Baseline, 12 weeks
Population: Analyzed was an intent-to-treat population using last observation carried forward as imputation technique. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 151 | 156
units on a scale | -2.58 (0.66) | -2.07 (0.66)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BAI score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.556, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-2.21 to 1.19]

11. Secondary Outcome: Correlation of Mean Changes From Baseline to 12 Week on the Adult ADHD Quality of Life-29 Total Score and of Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Investigator Rated:Screening Version Total Score
Description: AAQOL-29: Patient-reported outcome measure examining disease-specific functional impariments and quality of life for adults with ADHD. The domains included in the AAQOL are life productivity, psychological health, quality of relationships, and life outlook. Consistent with the majority of existing quality of life measures, higher scores on the AAQOL-29 indicate better functioning.
  CAARS-Inv:SV: Inattention subscale, Impulsivity subscale, and ADHD Index. Each item is scored on a 0 to 3 scale, assessing symptom severity over the past week. The total score is the sum of all subscale scores.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Number; unit: correlation coefficient
Arm/Group | Atomoxetine 20 - 50 mg BID and Placebo
Number analyzed (Participants) | 378
correlation coefficient | -0.591
Statistical Analysis 1: Comparison: Atomoxetine 20 - 50 mg BID and Placebo; Tested was the null hypothesis that AAQOL-29 total score and CAARS-Inv:SV total score are not correlated; Test type: Superiority or Other; p < 0.001, Pearson's Correlation Coefficient

12. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Habits Timeline Followback (TLFB) Incidence for Use of Alcohol
Description: Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of standard drinks that have been consumed.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: number of alcoholic drinks per day
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 119 | 121
number of alcoholic drinks per day | -0.21 (0.09) | -0.06 (0.09)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in TLFB incidence for use of alcohol score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.198, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.39 to 0.08]

13. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Habits Timeline Followback (TLFB) Incidence for Use of Caffeine
Description: Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of caffeine consumed by an individual. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: number of caffeinated drinks per day
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 162 | 163
number of caffeinated drinks per day | -0.23 (0.11) | -0.20 (0.11)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in TLFB incidence for use of caffeine score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.825, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.33 to 0.26]

14. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Habits Timeline Followback (TLFB) Incidence for Use of Drugs
Description: Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of recreational drugs other than marijuana an individual consumed and is expressed as the ratio of number of days on which drugs were used over the total number of days, resulting in a total score ranging from 0 to 1. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 2 | 2
ratio | 0.02 (0.01) | 0.02 (0.23)

15. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Habits Timeline Followback (TLFB) Incidence for Use of Nicotine
Description: Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. This subscale assesses the amount of nicotine consumed by an individual. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: number of nicotine products per day
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 70 | 70
number of nicotine products per day | 0.01 (0.51) | -0.81 (0.52)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in TLFB incidence for use of nicotine score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.233, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.53 to 2.17]

16. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Habits Timeline Followback (TLFB) Incidence for Use of Marijuana
Description: Variation of the Alcohol Timeline Followback (TLFB) which is a method for assessing the quantity of alcohol consumption on a daily basis. With a calendar as a guide, the interviewee provides a retrospective estimate of daily habits over a specified period of as long as the previous year. The goal is to provide a detailed record of patterns of use that can be used to guide treatment and to assess treatment outcome. Recorded is the number of joints that have been consumed.
Time Frame: Baseline, 12 weeks
Population: Analyzed was an intent-to-treat population using last observation carried forward technique. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: number of joints per day
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 26 | 20
number of joints per day | 0.09 (0.10) | 0.03 (0.12)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in TLFB incidence for use of marijuana score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.676, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.24 to 0.37]

17. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Fagerstrom Test for Nicotine Dependence (FTND)
Description: The FTND was designed to provide an ordinal measure of nicotine dependence related to cigarette smoking. It contains items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence. The FTND contains 4 yes-no and 2 multiple choice questions and can be used in a self-report format. The items on FTND are scored 0 to 3 for multiple choice items, the items are summed to yield a total score of 0-10 (0=minimum nicotine dependence; 10=maximum nicotine dependence).
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 48 | 42
units on a scale | 0.12 (0.25) | 0.43 (0.27)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in Fagerstorm Test for Nicotine Dependence score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.382, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.00 to 0.39]

18. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint on the Social Adaptation Self-Evaluation Scale (SASS)
Description: Patient completed scale that consists of 21 items that examine behavior and subjective perception, including satisfaction, self-perception and motivation in participating in and maintaining relationships with family and friends, satisfaction in work, home and leisure activities, and intellectual interests. Each item is scored from 0 to 3, corresponding to minimal and maximal social adjustment, with a total score range from 0 to 60.
Time Frame: Baseline, 12 weeks
Population: Analyzed was a intent-to-treat population using last observation carried forward imputation technique. Included were all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 165
units on a scale | 1.24 (0.39) | 1.46 (0.39)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in SASS score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.656, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.22, 95% CI 2-sided [-1.24 to 0.78]

19. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Driving Behavior Survey Self-Report
Description: 26 item self-rated driving survey with examples of driving behaviors, e.g.: putting on seat belt, driving within speed limits, yielding the right of way to other drivers. Items are rated on a 4-point scale (1 = not at all or rarely, 2 = sometimes, 3 = often, 4 = very often). The total score is the sum of the 26 items. A driving history is completed by self-report the first time a rater completes the Driving Behavior Survey (Self-Report). The total score ranges from 26 to 104.
Time Frame: Baseline, 12 weeks
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 140 | 142
units on a scale | 1.93 (0.98) | 3.54 (1.01)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in Driving Behavior Survey Self-Report score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.201, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -1.61, 95% CI 2-sided [-4.08 to 0.86]

20. Primary Outcome: Mean Change in the Conners' Adult ADHD Rating Scale-Investigator Rated: Screening Version (CAARS-Inv:SV) Total ADHD Symptom Score From Baseline to 12 Week Endpoint
Description: CAARS-Inv:SV is a 30-item scale containing 3 subscales: the Inattention subscale, the Hyperactivity-Impulsivity subscale, and the ADHD Index. The 18-item total ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each item is scored on a 0 to 3 scale (0=not at all, never; 1=just a little, once in a while; 2=pretty much, often; 3=very much, very frequently). The scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
Time Frame: Baseline, Week 12
Population: Intent-to-treat population was analyzed, including all randomized patients who had both a baseline and at least 1 post baseline score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 119 | 134
units on a scale | -14.88 (0.88) | -9.82 (0.85)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no difference in CAARS-Inv:SV score changes from baseline to 12-week endpoint between the atomoxetine group and the placebo group. With approximately 220 patients per arm, assuming a 68% completion rate and an estimated effect size of atomoxetine over placebo of 0.35, using a 5% significance level, the analysis was expected to have 90% power to detect a difference between atomoxetine and placebo at week 12; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Adjusted for treatment, investigator, visit, treatment-by-visit interaction, baseline score, baseline score-by-visit interaction; Mean Difference (Final Values) = -5.06, 95% CI 2-sided [-7.39 to -2.72]

21. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Driving Behavior Survey-Other Report
Description: 26-item driving survey completed by someone other than the patient/driver. Examples of driving behaviors included in the survey match those listed in the Self-Report version of the scale. Items are rated on a 4-point scale (1 = not at all or rarely, 2 = sometimes, 3 = often, 4 = very often). The total score is the sum of the 26 items and ranges from 26 to 104.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 13 | 11
units on a scale | 3.24 (3.67) | 2.63 (3.96)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in Driving Behavior Survey Other-Report score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.933, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = 0.61, 95% CI 2-sided [-16.41 to 17.63]

22. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Behavioral Regulation Section Score
Description: The BRIEF-A behavioral regulation subscale measures an individuals control over behavior in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 30 to 90.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -8.15 (0.83) | -5.20 (0.83)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Behavioral regulation score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.007, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -2.95, 95% CI 2-sided [-5.09 to -0.81]

23. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Emotional Control Section Score
Description: The BRIEF-A emotional control subscale assesses an individuals emotional control in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 10 to 30.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -1.98 (0.36) | -1.40 (0.36)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A emotional control section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.219, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-1.50 to 0.35]

24. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - GEC Section Score
Description: The BRIEF-A GEC rates the global executive composite of the patient in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 75 to 225.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -22.41 (1.86) | -14.83 (1.85)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A GEC section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -7.58, 95% CI 2-sided [-12.37 to -2.78]

25. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Inconsistency Section
Description: The BRIEF-A Inconsistency rates the behavioral inconsistency displayed by the patient in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 0 to 20.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -0.51 (0.15) | -0.42 (0.15)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Inconsistency section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.644, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.47 to 0.29]

26. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Infrequency Section
Description: Standardized measure assessing adult executive functioning/self-regulation in his/her everyday environment. Extent to which respondent answers additional items in an unusual and infrequent direction. Form is designed to be completed by adults 18-90 years of age, including adults with wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. Total score ranges from 0 to 5.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | 0.27 (0.05) | 0.16 (0.05)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEFS-A infrequency score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.097, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.02 to 0.25]

27. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Inhibit Section
Description: The BRIEF-A Inhibit rates an individual's inhibition in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -2.62 (0.23) | -1.65 (0.23)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Inhibit Section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.97, 95% CI 2-sided [-1.57 to -0.37]

28. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Initiate Section
Description: The BRIEF-A Initiate rates an individual's initiative behaviors in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -2.41 (0.25) | -1.74 (0.25)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Initiate section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.044, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.33 to -0.02]

29. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Metacognition Section
Description: BRIEF-A Metacognition subscale is a standardized measure assessing individual's ability to systematically solve problems via planning and organization while sustaining these task-completion efforts in active working memory. Form is designed to be completed by adults, including adults with wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior never observed, 2=behavior sometimes observed, and 3=behavior often observed - higher ratings indicate greater perceived impairment. Total score ranges from 40 to 120.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -14.13 (1.14) | -9.64 (1.13)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Metacognition section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -4.49, 95% CI 2-sided [-7.43 to -1.55]

30. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Negativity Section
Description: The BRIEF-A Negativity asseses an indivduals' perceived negativity in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 0 to 10.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -0.85 (0.14) | -0.71 (0.14)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A negativity section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.456, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.51 to 0.23]

31. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Organization of Materials Section
Description: The BRIEF-A Organization of Materials assesses an individuals' organizing skills in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -2.50 (0.25) | -1.85 (0.25)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Organization of Materials section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.051, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-1.31 to 0.00]

32. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Plan/Organize Section
Description: The BRIEF-A Plan/Organize asseses an individuals' capabilities to plan and organize in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Behavior is rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 10 to 30.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -3.62 (0.33) | -2.28 (0.33)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Plan/Organize section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.002, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.19 to -0.47]

33. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - SHIFT Section
Description: The BRIEF-A Shift assess an individuals' shifting between different behaviors in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -1.49 (0.20) | -0.96 (0.20)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A SHIFT section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.045, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-1.04 to -0.01]

34. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Self Monitor Section
Description: The BRIEF-A Self Monitor assesses an individuals' capacity to self monitor in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -2.03 (0.20) | -1.20 (0.20)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Self Monitor Section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.001, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.35 to -0.32]

35. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Task Monitor Section
Description: The BRIEF-A Task Monitor assesses an individuals's ability to monitor a task in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 6 to 18.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -2.28 (0.20) | -1.57 (0.20)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Task Monitor section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.008, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.23 to -0.19]

36. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Behavior Rating Inventory of Executive Function-Adult Version Self Report (BRIEF-A) - Working Memory Section
Description: The BRIEF-A Working Memory assesses an individuals' memory function in his or her everyday environment. The self-report form is designed to be completed by adults 18-90 years of age, including adults with a wide variety of developmental, systemic, neurological, and psychiatric disorders. Observations are rated on a 3-point Likert scale, with 1=behavior is never observed, 2=behavior is sometimes observed, and 3=behavior is often observed - higher ratings indicate greater perceived impairment. The total score ranges from 8 to 24.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 161 | 167
units on a scale | -3.48 (0.26) | -2.18 (0.26)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in BRIEF-A Working Memory section score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-1.98 to -0.63]

37. Secondary Outcome: Mean Change From Baseline to 12-Week Endpoint on the Epworth Sleepiness Scale (ESS)
Description: Used to determine the level of daytime sleepiness. The ESS is a self-rated questionnaire with 8 items that describe normative daily situations known to vary in their soporific qualities. Subjects rate the likelihood of dozing off or falling asleep in each of these situations. Each item is rated on a 4-point scale from 0 (would never doze) to 3 (high chance of dozing). The item scores are summed to produce a total score (range of 0-24). Score >10 (95th percentile) are considered to be suggestive of significant daytime sleepiness.
Time Frame: Baseline, 12 weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 187 | 196
units on a scale | -1.76 (0.29) | -1.07 (0.28)
Statistical Analysis 1: Comparison: Atomoxetine vs Placebo; Tested was the null hypothesis that there is no statistically significant difference in ESS score changes from baseline to 12-week endpoint between atomoxetine and placebo treatment groups; Test type: Superiority or Other; p = 0.065, ANCOVA; ANCOVA model with terms for baseline score, treatment, and investigator; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-1.42 to 0.04]

38. Secondary Outcome: Responders by Baseline Smoking Status
Description: Baseline smoking status was recorded and associations to response to treatment were determined. Response was defined as 25% or greater decrease in ADHD symptoms as measured by the CAARS-Inv:SV total ADHD symptom score. The 18-item total CAARS-Inv:SV ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each item is scored on a 0 to 3 scale (0=not at all, never; 1=just a little, once in a while; 2=pretty much, often; 3=very much, very frequently). The scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Atomoxetine 20 - 50 mg BID, Smokers | Atomoxetine 20 - 50 mg BID, Non-smokers | Placebo, Smokers | Placebo Non-smokers
Number analyzed (Participants) | 91 | 128 | 94 | 131
participants | 54 | 60 | 29 | 53
Statistical Analysis 1: Comparison: Atomoxetine 20 - 50 mg BID, Smokers vs Atomoxetine 20 - 50 mg BID, Non-smokers vs Placebo, Smokers vs Placebo Non-smokers; Tested was the null hypothesis that smoking status is not a predictor of response to atomoxetine treatment compared with placebo; Test type: Superiority or Other; p = 0.788, Cochran-Mantel-Haenszel; Tested was smoking status across treatment

39. Secondary Outcome: Strong Responders by Baseline Smoking Status
Description: Baseline smoking status was recorded and associations to response to treatment were determined. Strong response was defined as 40% or greater decrease in ADHD symptoms as measured by the CAARS-Inv:SV total ADHD symptom score. The 18-item total CAARS-Inv:SV ADHD symptom score is the sum of the Inattention and Hyperactivity-Impulsivity subscales. Each item is scored on a 0 to 3 scale (0=not at all, never; 1=just a little, once in a while; 2=pretty much, often; 3=very much, very frequently). The scale assesses symptom severity over the past week. The total score ranges from 0 to 54.
Time Frame: 12 weeks
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Atomoxetine 20 - 50 mg BID, Smokers | Atomoxetine 20 - 50 mg BID, Non-Smokers | Placebo, Smokers | Placebo, Non-Smokers
Number analyzed (Participants) | 91 | 128 | 94 | 131
participants | 38 | 41 | 19 | 31
Statistical Analysis 1: Comparison: Atomoxetine 20 - 50 mg BID, Smokers vs Atomoxetine 20 - 50 mg BID, Non-Smokers vs Placebo, Smokers vs Placebo, Non-Smokers; Tested was the null hypothesis that smoking status is not a predictor of strong response to atomoxetine treatment compared with placebo; Test type: Superiority or Other; p = 0.482, Cochran-Mantel-Haenszel — Tested was smoking status across treatment

ADVERSE EVENTS:
Arm/Group | Atomoxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/220 | 1/225
Other Adverse Events (participants affected / at risk) | 147/220 | 121/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=220) | Placebo (N=225)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=220) | Placebo (N=225)
Abdominal discomfort (Gastrointestinal disorders) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 19 (19) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 11 (12) | 2 (2)
Nausea (Gastrointestinal disorders) | 31 (35) | 11 (11)
Vomiting (Gastrointestinal disorders) | 7 (7) | 7 (7)
Fatigue (General disorders) | 13 (13) | 13 (14)
Irritability (General disorders) | 12 (13) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (6) | 10 (10)
Pharyngitis streptococcal (Infections and infestations) | 5 (5) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 13 (13)
Weight decreased (Investigations) | 7 (7) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 27 (27) | 5 (5)
Dizziness (Nervous system disorders) | 11 (11) | 3 (3)
Headache (Nervous system disorders) | 13 (15) | 18 (19)
Sedation (Nervous system disorders) | 6 (7) | 3 (3)
Somnolence (Nervous system disorders) | 10 (10) | 4 (4)
Abnormal dreams (Psychiatric disorders) | 6 (6) | 8 (8)
Anxiety (Psychiatric disorders) | 9 (10) | 5 (5)
Insomnia (Psychiatric disorders) | 23 (23) | 10 (10)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days